CLINICAL TRIAL: NCT06288659
Title: Aneurysmal Subarachnoid Hemorrhage Treatment Based on Intraventricular Intracranial Pressure Monitoring: A Prospective, Multicenter, Randomized and Controlled Trial
Brief Title: aSAH Treatment Based on Intraventricular ICP Monitoring: A Prospective, Multicenter, Randomized and Controlled Trial
Acronym: ASTIM-MT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhu, Vice director of neurosurgery department, Huashan Hospital, Fudan University, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2024-050
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Intracranial Pressure Increase
Keywords: Aneurysmal subarachnoid hemorrhage; Intraventricular intracranial pressure monitoring; Multicenter randomized clinical trail
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aSAH treatment based on Intraventricular ICP monitoring (Experimental): In the acute phase of aSAH (following endovascular or craniotomy occlusion of the aneurysm), a ventricular ICP monitoring probe is surgically implanted. And the postoperative management of ICP is guided by quantifiable ICP parameters. The remaining treatments are consistent with those in the control group.
  Interventions: Device: Intraventricular intracranial pressure monitoring
- aSAH treatment without Intraventricular ICP monitoring (No Intervention): Only aSAH treatment surgery is performed without intraventricular ICP monitoring probe implantation. The treatment is not guided by ICP monitoring, and instead, aSAH treatment is conducted based on clinical signs and CT imaging to assess ICP.

INTERVENTIONS:
Device: Intraventricular intracranial pressure monitoring — The postoperative management of ICP is guided by quantifiable Intraventricular ICP parameters. The remaining treatments are consistent with those in the control group.
  Arms: aSAH treatment based on Intraventricular ICP monitoring

SUMMARY:
ASTIM is a multicenter, prospective, randomised, blinded end-point assessed trial, to investigate the efficacy and safety of treatment based on intracranial pressure monitoring in improving the prognosis of patients with aneurysmal subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) is a severe type of cerebral hemorrhage, characterized by a high mortality and disability rate, approximately 85% of SAH cases are attributed to ruptured intracranial aneurysms (RIAs), which is called aneurysmal SAH (aSAH). Improving the prognosis of patients with aSAH has become a pressing and significant issue.

The rupture of an aneurysm results in a significant amount of blood entering the subarachnoid space, triggering an increase in intracranial pressure (ICP). This escalated ICP, coupled with the compression from the hematoma, severely impairs brain tissue function, leading to a cascade of irreversible neurological impairments, such as abnormal blood pressure, respiratory arrest, and cardiac arrest. Systematic reviews and meta-analysis found that the incidence rate of elevated ICP (ICP > 20mmHg) in post-aSAH patients was 70.69%, with higher levels (according to the Hunt-Hess scale, WFNS scale, or modified Fisher grade) being more prevalent for increased ICP.

The utilization of Intraventricular ICP monitoring in patients with aSAH offers the advantage of obtaining real-time, accurate data on intracranial pressure, enabling more precise and timely control of cranial pressure. However, there is a dearth of high-level randomized controlled trial evidence supporting the use of ICP in the treatment of aSAH. Given the potential utility of ICP monitoring in aSAH management and its current lack of high-level evidence in evidence-based medicine, we intend to pursue the research.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of aSAH: presence of SAH symptoms, confirmed by CT scan or lumbar puncture. CTA or DSA confirms ruptured intracranial aneurysm (IA) as the cause. Decision made to perform craniotomy clipping or endovascular treatment within 72 hours aiming for a single procedure to cure the bleeding artery aneurysm;
* Age ≥ 18 years;
* The onset of symptoms should occur within 72 hours;
* The Hunt-Hess grade is between 2 and 4, and the CT imaging findings correspond to a modified Fisher grade of 2 to 4.
* Obtain the consent of the patient and their family members, and have them sign an informed consent form.

Exclusion Criteria:

* Pregnancy or lactation period;
* Patients presenting with bilateral dilated pupils upon admission;
* Patients with concurrent tumors, hemorrhagic diseases, or other severe underlying conditions (such as chronic obstructive pulmonary disease, multiple organ dysfunction syndrome, severe diabetes mellitus, congestive heart failure, and chronic kidney disease);
* Patients with a history of brain disorders or previous brain surgeries;
* Hemorrhage attributable to causes other than aneurysm;
* Aneurysmal rupture bleeding concurrent with moyamoya disease;
* Other underlying conditions that impact prognosis;
* Patients volunteering for ICP monitoring;
* Participants in other ongoing clinical trails;
* Other circumstances deemed inappropriate for inclusion (to be determined by two physicians).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The rate of good neurological functional prognosis | 90 days
  The proportion of patients with modified Rankin Scale (mRS) scores 0-2. The mRS is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability. A mRS ≤ 2 indicated a good clinical outcome, and a mRS 5-6 indicated a poor clinical outcome.

SECONDARY OUTCOMES:
The rate of good neurological functional prognosis | 30 days, 180days
  Proportion of patients with modified Rankin Scale (mRS) scores 0-2
The rate of good prognosis by Glasgow Outcome Scale-Extended (GOS-E) | 30 days, 90 days, 180days
  The GOS-E is an ordinal hierarchical scale ranging from 1 to 8, with lower scores indicating more severe disability.
Mortality | 30 days, 90 days, 180days
  Proportion of patients who died.
Incidence of VP shunt-related hydrocephalus | 90 days
  Incidence of hydrocephalus requiring ventriculoperitoneal shunt within 90days.
Incidence of Delayed Cerebral Ischemia | 90 days
  Proportion of delayed cerebral ischemia occurring within 90 days.
Incidence of epilepsy | 90 days
  Proportion of symptomatic epilepsy occurring within 90 days.

OTHER OUTCOMES:
Incidence of intracranial infection | 90 days
  The cerebrospinal fluid culture demonstrates positive findings for pathogenic bacteria, or the cerebrospinal fluid exhibits an elevated count of more than 1000 white blood cells with a predominance of polymorphonuclear cells, accompanied by decreased glucose levels and increased lactate levels in the cerebrospinal fluid.
Incidence of bleeding from puncture site | 90 days
  This refers to intracranial bleeding resulting from ventricular puncture, which can be confirmed via a head CT scan.
Incidence of poor healing in surgical incisions | 90 days
  This encompasses infection and suppuration at the ICP incision site, potentially impeding proper wound closure.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhu, Ph.D., Principal Investigator — Department of Neurosurgery, Huashan Hospital, Fudan University; Xuehai Wu, Ph.D., Principal Investigator — Department of Neurosurgery, Huashan Hospital, Fudan University
Locations (1):
- Department of Neurosurgery, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macdonald RL, Schweizer TA. Spontaneous subarachnoid haemorrhage. Lancet. 2017 Feb 11;389(10069):655-666. doi: 10.1016/S0140-6736(16)30668-7. Epub 2016 Sep 13. PMID 27637674
- [Background] Etminan N, Chang HS, Hackenberg K, de Rooij NK, Vergouwen MDI, Rinkel GJE, Algra A. Worldwide Incidence of Aneurysmal Subarachnoid Hemorrhage According to Region, Time Period, Blood Pressure, and Smoking Prevalence in the Population: A Systematic Review and Meta-analysis. JAMA Neurol. 2019 May 1;76(5):588-597. doi: 10.1001/jamaneurol.2019.0006. PMID 30659573
- [Background] Neifert SN, Chapman EK, Martini ML, Shuman WH, Schupper AJ, Oermann EK, Mocco J, Macdonald RL. Aneurysmal Subarachnoid Hemorrhage: the Last Decade. Transl Stroke Res. 2021 Jun;12(3):428-446. doi: 10.1007/s12975-020-00867-0. Epub 2020 Oct 19. PMID 33078345
- [Background] Ironside N, Buell TJ, Chen CJ, Kumar JS, Paisan GM, Sokolowski JD, Liu KC, Ding D. High-Grade Aneurysmal Subarachnoid Hemorrhage: Predictors of Functional Outcome. World Neurosurg. 2019 May;125:e723-e728. doi: 10.1016/j.wneu.2019.01.162. Epub 2019 Feb 6. PMID 30735864
- [Background] Seule M, Oswald D, Muroi C, Brandi G, Keller E. Outcome, Return to Work and Health-Related Costs After Aneurysmal Subarachnoid Hemorrhage. Neurocrit Care. 2020 Aug;33(1):49-57. doi: 10.1007/s12028-019-00905-2. PMID 31919809
- [Background] Hoh BL, Ko NU, Amin-Hanjani S, Chou SH-Y, Cruz-Flores S, Dangayach NS, Derdeyn CP, Du R, Hanggi D, Hetts SW, Ifejika NL, Johnson R, Keigher KM, Leslie-Mazwi TM, Lucke-Wold B, Rabinstein AA, Robicsek SA, Stapleton CJ, Suarez JI, Tjoumakaris SI, Welch BG. 2023 Guideline for the Management of Patients With Aneurysmal Subarachnoid Hemorrhage: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2023 Jul;54(7):e314-e370. doi: 10.1161/STR.0000000000000436. Epub 2023 May 22. PMID 37212182
- [Background] Heuer GG, Smith MJ, Elliott JP, Winn HR, LeRoux PD. Relationship between intracranial pressure and other clinical variables in patients with aneurysmal subarachnoid hemorrhage. J Neurosurg. 2004 Sep;101(3):408-16. doi: 10.3171/jns.2004.101.3.0408. PMID 15352597
- [Background] Robba C, Graziano F, Rebora P, Elli F, Giussani C, Oddo M, Meyfroidt G, Helbok R, Taccone FS, Prisco L, Vincent JL, Suarez JI, Stocchetti N, Citerio G; SYNAPSE-ICU Investigators. Intracranial pressure monitoring in patients with acute brain injury in the intensive care unit (SYNAPSE-ICU): an international, prospective observational cohort study. Lancet Neurol. 2021 Jul;20(7):548-558. doi: 10.1016/S1474-4422(21)00138-1. PMID 34146513